CLINICAL TRIAL: NCT07170189
Title: A Phase 1, Open-label, Randomized, Five-Part Study to Assess the Pharmacokinetics and Safety of Tablet and Capsule Formulations of HU6 in Overweight Participants.
Brief Title: Phase 1, Open-Label, Randomized, Study of the Safety and Pharmacokinetics of HU6
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RIV-HU6-108
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Experimental: Active Treatment HU6 450 mg tablet (Experimental): Drug: HU6 450 mg single tablet once daily (QD)
  Interventions: Drug: HU6
- Experimental: Active Treatment HU6 150 mg x 3 tablets (Experimental): Drug: HU6 150 mg x 3 tablets QD
  Interventions: Drug: HU6
- Experimental: Active Treatment HU6 (150 mg tablet × 2) BID (Experimental): Drug: HU6 300 mg dose (supplied as HU6 150 mg tablet × 2) BID (q12 hours)
  Interventions: Drug: HU6
- Experimental: Active Treatment HU6 150 mg drug substance in a capsule × 3 (450 mg total) (Experimental): Drug: HU6 150 mg drug substance in a capsule × 3 (450 mg total dose) QD
  Interventions: Drug: HU6
- Experimental: Active Treatment HU6 150 mg granulated blend in a capsule × 3 (450 mg total) (Experimental): Drug: HU6 150 mg granulated blend in a capsule × 3 (450 mg total dose) QD
  Interventions: Drug: HU6

INTERVENTIONS:
Drug: HU6 — HU6 tablet or capsule

SUMMARY:
This is a five-part study being conducted to evaluate the safety, tolerability and pharmacokinetics of the HU6 tablet and capsule formulations at steady state in the fed and fasted state for HU6 450 mg once daily (QD) dose (as single or multiple tablets) or HU6 300 mg twice daily (BID) (supplied as two 150 mg tablets) or HU6 150 mg drug substance in a capsule × 3 (450 mg total dose) QD or HU6 150 mg granulated blend in a capsule × 3 (450 mg total dose) QD.

DETAILED DESCRIPTION:
This is a five-part study being conducted to evaluate the safety, tolerability and pharmacokinetics of the HU6 tablet and capsule formulations at steady state in the fed and fasted state for 450 mg once daily (QD) dose (as single or multiple tablets) or 300 mg twice daily (BID) (supplied as two 150 mg tablets) or HU6 150 mg drug substance in a capsule × 3 (450 mg total dose) QD or HU6 150 mg granulated blend in a capsule × 3 (450 mg total dose) QD. Population pharmacokinetic (popPK) modeling indicated a potential difference in PK profile when multiple dose units are administered versus a single dose unit in tablet and capsule formulations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age at time of signing the informed consent.
* Body mass index (BMI) ≥ 25 kg/m2 at Screening.
* Medically stable in the opinion of the investigator based on medical history, physical examination, vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and general observations. Note that Screening abnormalities or findings outside the normal ranges for any clinical assessments that are considered clinically significant by the Investigator (clinical laboratory tests, ECG, vital signs) may be repeated once at the discretion of the Investigator(s), and results that continue to be outside the normal ranges must be judged by the investigator to be not clinically significant and acceptable for study participation.
* Signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this clinical protocol.

Exclusion Criteria:

* Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease as determined by the investigator and if deemed necessary, in consultation with the medical monitor, which may impact safety.
* History of cancer (except for treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening.
* Any surgical or medical condition or history that, in the opinion of the investigator, and if deemed necessary, in consultation with the medical monitor, may potentially alter the absorption, metabolism, or excretion of IMP, such as, but not limited to, gastric bypass surgery or gallbladder removal surgery or significant small bowel resections.
* Contraindication to IMP or its excipients and/or history of anaphylactic reactions or clinically significant allergic reaction.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2025-10-13 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
b. To estimate multiple dose plasma pharmacokinetics of HU6 with emphasis on the exposure parameter of maximum concentration (Cmax). | 28 days
  To estimate multiple dose plasma pharmacokinetics of HU6 with emphasis on exposure parameters of maximum concentration (Cmax), after multiple dose administration of the tablet and capsule formulations of HU6

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No